CLINICAL TRIAL: NCT00664807
Title: Medtronic Genetic Arrhythmia Markers for Early Detection
Brief Title: Medtronic Genetic Arrhythmia Markers for Early Detection (GAME Study)
Acronym: GAME
Status: Completed | Type: Observational
Sponsor: Medtronic Corporate Technologies and New Ventures (Industry)
Responsible Party: Tara Nahey/Senior Scientist, Medtronic Corporate Technologies and New Ventures
Other Study IDs: MDT-CTNV-001
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia; Atrial Fibrillation; Sick Sinus Syndrome
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia; Atrial Fibrillation; Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To generate a list of potential genetic markers that correlate with an increased risk of life-threatening arrhythmias.

To evaluate ECG-based risk markers such as heart rate variability and T-wave Alternans for their association with arrhythmic events.

DETAILED DESCRIPTION:
The primary objective is to establish the role of genetics in life-threatening arrhythmias leading to sudden cardiac death (SCD) and the potential utility of genetic markers in risk stratification of patients to receive an implantable cardiac defibrillator (ICD). The successful accomplishment of this goal would serve as the basis for future work on a specific diagnostic test that can be used to assess risks of threatening arrhythmias in order to quality patients for implantation of an ICD.

* to identify single nucleotide polymorphisms (SNPs) that can be used to identify individuals in need of an ICD.

The secondary objectives involve more detailed analysis to search for potentially unidentified genetic markers of risk for SCD.

1. to identify genes associated with SCD susceptibility.
2. to identify risk factors associated with SCD as found in the case report form (CRF).
3. to correlate SNPs with co-morbidities in the subjects as found in the CRF information.
4. to study the association between parameters derived from Holter recordings and predictors of life-threatening arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

The following criteria apply to all subjects:

* Subject has an ICD or CRT ICD implanted
* Subject must be on optimal medical therapy
* Subject is a Caucasian with all 4 grandparents believed to be Caucasian
* Subject has had a myocardial infarction (MI) prior to ICD implantation
* Subject is willing and able to comply with the study protocol
* Subject is willing and able to sign and date the study Informed Consent and HIPAA Authorization (US)

Case Inclusion Criteria:

The following criteria apply to case subjects only:

* Subject is at least 40 years of age at time of ICD implantation
* Subject has at least one documented life-threatening arrhythmia (LTA) on their ICD that can transferred as a save-to-disk or has had an LTA documented in their medical history. LTA is defined as a true VT/VF episode with cycle length less than or equal to 400ms that was terminated by the device.

Control Inclusion Criteria:

The following criteria apply to control subjects only:

* Subject is currently at least 70 years of age
* Subject has haad currently implanted Medronic ICD for a minimum of three years

Exclusion Criteria:

The following criteria apply to all subjects:

* Subject has received a bone marrow or heart transplant at any time
* Subject has a previously identified cause for arrhythmias (Brugada, LQT, HCM)

Control Exclusion Criteria:

The following criteria apply to control subjects only:

* Subject has had a potentially LTA documented on their ICD
* Subject was previously identified as having a LTD at any time in life
* Subject has had the memory on their ICD cleared at any time in the past three years.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic, Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of single nucleotide polymorphisms as predictors of life-threatening arrhythmias. | one year

SECONDARY OUTCOMES:
Positive predictive value of genetic markers as predictors of life-threatening arrhythmias. | one year
Association between risk factors identified in the CRF and life-threatening arrhythmias. | one year
Correlation of SNPs to other co-morbidities identified in the CRF information. | one year
Association between ECG-based risk markers and life-threatening arrhythmias. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, M.D., Principal Investigator — Scripps Translational Science Institute, La Jolla, CA USA; Robert Kowal, M.D.,Ph.D., Principal Investigator — HeartPlace Baylor, Dallas, TX USA
Locations (1):
- Arkansas Cardiology, PA, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Murray SS, Smith EN, Villarasa N, Nahey T, Lande J, Goldberg H, Shaw M, Rosenthal L, Ramza B, Alaeddini J, Han X, Damani S, Soykan O, Kowal RC, Topol EJ; GAME Investigators. Genome-wide association of implantable cardioverter-defibrillator activation with life-threatening arrhythmias. PLoS One. 2012;7(1):e25387. doi: 10.1371/journal.pone.0025387. Epub 2012 Jan 11. PMID 22247754